CLINICAL TRIAL: NCT05789589
Title: A Phase I/II Study to Assess Safety and Preliminary Evidence of a Therapeutic Effect of Azeliragon Combined With Stereotactic Radiation Therapy in Patients With Brain Metastases
Brief Title: Effect of Azeliragon Combined With Stereotactic Radiation Therapy in Patients With Brain Metastases
Acronym: ADORATION
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Collaborators: Miami Cancer Institute (Other); Cantex Pharmaceuticals Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2022-KOT-002
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Metastasis; Metastatic Cancer; Brain Metastases; Brain Metastases, Adult
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Brain Neoplasms | interventions — azeliragon; Radiosurgery; Adrenal Cortex Hormones; Dexamethasone; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Azeliragon and Stereotactic Radiosurgery (SRS) (Experimental): In the Phase 1 portion of the study, three treatment regimens will be systematically evaluated:
  1. Azeliragon + SRS + loading corticosteroid dose (LD) + corticosteroid taper (CT)
  2. Azeliragon + SRS + loading corticosteroid dose (LD)
  3. Azeliragon + SRS
  The starting cohort will receive Regimen #2, and depending on the tolerability, participants will be allocated to subsequent cohorts as follows: if Regimen #2 is not well tolerated, participants will be allocated to Regimen #1; if #2 is well tolerated, participants will be allocated to Regimen #3.
  Once a Regimen has been identified as safe and tolerable, it will be used for the Phase 2 portion of the study.
  Interventions: Drug: Azeliragon; Radiation: Stereotactic radiosurgery; Drug: Corticosteroid

INTERVENTIONS:
Drug: Azeliragon — Dosing will begin on Day 0 with the loading dose and continue daily through Day 7. Starting on Day 8, dosing will resume with the continuous dose until disease progression or 8 weeks. If there is evidence of antitumor effect at 8 weeks, dosing may continue for up 2 two years.
  All doses are taken orally. There are three levels of dosing, including a starting dose and two lower levels of dosing. Participants will start with the starting dose, and in the event of the dose limiting toxicities, the dose will be reduced as described below.
  Starting Dose Level: 30 mg twice daily (Loading Dose) or 20 mg once daily (Continuous Dose) Dose Level -1: 15 mg twice daily (Loading Dose) or 10 mg once daily (Continuous Dose) Dose Level -2: 15 mg once daily (Loading Dose) or 5 mg once daily (Continuous Dose)
  Other Names: TTP488; PF-04494700
Radiation: Stereotactic radiosurgery — Patients will undergo standard of care SRS as per the treating facility's policies.
Drug: Corticosteroid — Two corticosteroid regimens are used depending on the study cohort. Cohorts 1 and 2 will receive the loading dose (LD). Only Cohort 1 will receive the corticosteroid taper (CT).
  LD: Oral (8 mg) or IV bolus dose (10 mg) of dexamethasone or 40 to 80 mg of methylprednisolone on the day of SRS CT: Oral 2-4 mg of dexamethasone twice daily for 5 days and then 2-4 mg daily for 5 days at the discretion of the treating physician (concurrent use of a proton pump inhibitor or H2 receptor antagonists are encouraged during the CT).
  Other Names: dexamethasone; methylprednisolone

SUMMARY:
To determine the safety and efficacy of using the drug azeliragon combined with stereotactic radiosurgery. Specifically, to determine if this combination will lead to improved response in the brain (tumor shrinking in size) and overall tumor control (how long tumor remains controlled).

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have histologically or cytologically confirmed diagnosis of cancer within the past 5 years. If original histologic proof of malignancy is > 5 years, then biological [such as presence of tumor markers, circulating tumor (ctDNA), etc.], or pathological (i.e., more recent) confirmation is required (e.g., from a systemic metastasis or brain metastasis)
2. Age ≥ 18
3. Karnofsky performance status ≥ 50 or Eastern Cooperative Oncology Group (ECOG) ≤ 3
4. Brain metastasis with a maximum tumor diameter of the largest lesion ≤ 2 cm
5. Patients must have discontinued corticosteroids at least 5 days prior to SRS. (Note: This does not apply to corticosteroids administered as part of this protocol.)
6. Patients must not be pregnant (positive pregnancy test) or breast feeding. Effective contraception (men and women) must be used in patients of child-bearing potential during radiotherapy and for 6 months after.
7. Patients who have received prior SRS are eligible, provided that there are new non-irradiated brain lesions and that the patient is ≥ 2 months post prior cranial radiation therapy
8. Patient has adequate biological parameters as demonstrated by the following blood counts at Screening (obtained ≤ 14 days prior to enrollment):

   * Absolute neutrophil count (ANC) ≥ 1.0 × 10^9/L
   * Platelet count ≥ 75,000/mm^3 (75 × 10^9/L)
   * Hemoglobin (Hgb) ≥ 9 g/dL without transfusion or growth factor support
9. Absolute neutrophil count (ANC) ≥ 1.0 × 10^9/L; Platelet count ≥ 75,000/mm^3 (75 × 10^9/L); Hemoglobin (Hgb) ≥ 9 g/dL without transfusion or growth factor support
10. Patient has the following blood chemistry levels at Screening (obtained ≤ 14 days prior to enrollment):

    * Aspartate aminotransferase (AST; SGOT), alanine transaminase (ALT; SGPT) ≤ 2.5 × upper limit of normal range (ULN). Total bilirubin ≤ 1.5 × ULN.
    * Estimated creatinine clearance of > 60 mL/min (per Cockcroft-Gault formula)

Exclusion Criteria:

1. Patients with leptomeningeal disease
2. Patients unable to undergo magnetic resonance imaging (MRI)
3. Patients receiving Cytochrome P450 (CYP) 2C8 inhibitors as indicated in the protocol
4. Patients with a gastrointestinal condition that could interfere with swallowing or absorption.
5. Females of childbearing potential who are sexually active or males with female partners of childbearing potential, where either the female or the male is unwilling to use a highly effective method of contraception during the trial and for 6 months after the last administration of azeliragon.
6. Patients with concurrent participation in another interventional clinical trial or use of another investigational agent within 7 days of starting azeliragon. Patients who are participating in non-interventional clinical trials (e.g., QOL, imaging, observational, follow-up studies, etc.) are eligible, regardless of the timing of participation.
7. Any patient that in the opinion of the principal investigator is not an appropriate candidate for this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2027-03-16 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Total Dose-Limiting Toxicities (DLTs) | 4 weeks
  A DLT of the azeliragon and corticosteroid regimen is defined as any central nervous system (CNS)-specific Grade ≥ 2 toxicity requiring corticosteroid treatment or any Grade ≥ 3 events that are not clearly due to the underlying disease or extraneous causes. DLTs will be considered up to four weeks after SRS.

SECONDARY OUTCOMES:
CNS treatment-related adverse events | 24 months
  Participants are evaluated for treatment-related adverse events (AEs). The total count of treatment-related AEs for all participants and those specifically in the central nervous system will be calculated. CNS treatment-related adverse events will be reported as percent of total treatment-related AEs.
Early brain metastases response rate | 8 weeks
  Response and progression will be evaluated using the Response Assessment in Neuro-Oncology (RANO) criteria for brain metastasis (RANO-BM). The percent of patients with a complete response (CR) or partial response (PR) will be categorized individually and then together will be used to compare to the historical comparator of 24% with SRS alone.
Intracranial objective response rate | 6 months
  Response and progression will be evaluated using RANO-BM. The percent of patients with CR, PR, or stable disease (SD) will be calculated.
Intracranial objective response rate | 12 months
  Response and progression will be evaluated using RANO-BM. The percent of patients with CR, PR, or SD will be calculated.
Lesion-specific local tumor control rate | 6 months
  Local failure will be defined using the following criteria: For lesions measuring more than 5 mm in the baseline (volumetric) scan: At least 50% increase in the product of the two largest perpendicular diameters (compared to the smallest product measured for the same lesion). For lesions measuring 5 mm or less in the baseline (volumetric) scan: At least 100% increase in the product of the two largest perpendicular diameters (compared to the smallest product measured for the same lesion). Radiation necrosis will not be considered tumor progression.
  Lesion-specific tumor control rate is defined as the percent of lesions that do not meet criteria for local failure as defined above.
Lesion-specific local tumor control rate | 12 months
  Local failure will be defined using the following criteria: For lesions measuring more than 5 mm in the baseline (volumetric) scan: At least 50% increase in the product of the two largest perpendicular diameters (compared to the smallest product measured for the same lesion). For lesions measuring 5 mm or less in the baseline (volumetric) scan: At least 100% increase in the product of the two largest perpendicular diameters (compared to the smallest product measured for the same lesion). Radiation necrosis will not be considered tumor progression.
  Lesion-specific tumor control rate is defined as the percent of lesions that do not meet criteria for local failure as defined above.
Neurocognitive outcomes battery | 24 months
  The following tests are included:
  * Hopkins Verbal Learning Test (HVLT)
  * Controlled Oral Word Association Test (COWAT)
  * Trail Making Test Part A
  * Trail Making Test Part B
  * Grooved Pegboard
  HVLT raw scores are derived for Total Recall, Delayed Recall, and Retention (% retained). COWAT is measured by summing the number of acceptable words produced for three separate letters during one minute each. The trail making tests are measured by the time they take to complete. The grooved pegboard is scored by the amount of time it takes to place the pegs correctly in the pegboard. Higher scores on HVLT and COWAT and faster times on the trail making and pegboard indicate better neurocognitive function. All tests are then standardized based on published norms and transformed so that higher values represent improved cognition.
  The endpoint is defined as a decline of greater than 1 standard deviation from baseline on at least 1 of the 5 neurocognitive tests.
Change in patient-reported outcomes (PROs) | Baseline to 24 months
  PROs will be assessed using the MD Anderson Symptom Inventory for brain tumors (MDASI-BT), a validated assessment in people with brain metastases. It is a 28-item questionnaire that includes 13 symptom severity items, 6 symptom interference items, and 9 brain-tumor specific symptom items. Experience of each item "in the last 24 hours" is rated on a 10-point Likert scale where a higher score indicates worse outcomes.
  Ratings are averaged into several subscale scores: mean core symptom severity, mean brain tumor symptom severity, and mean interference. The change score from baseline to 24 months will be calculated by subtracting the 12-month overall score from the baseline overall score. Positive values indicate improved outcomes and negative values indicate worse outcomes.
Change in quality of life (QOL) using EORTC QLQ-C30 | Baseline to 24 months
  European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 consists of 30 items and measures an individual's functioning and symptoms for all cancer types. Questions are grouped into 5 multi-item functional scales; 3 multi-item symptom scales; a 2-item global health status scale; 5 single items assessing additional symptoms commonly reported by cancer patients, and 1 item on the financial impact of the disease.
  Raw QLQ-C30 scores are transformed to standardized scores (0 to 100); a higher score represents a better level of functioning or a worse level of symptoms. A Summary Score is calculated from the mean of 13 of the 15 scales (excluding Global Quality of Life and Financial Impact scales). The symptom scales are reversed to obtain uniform direction of all scales.
  The change score from baseline to 24 months will be calculated by subtracting the 24-month score from the baseline score. Negative values indicate improved QOL.
Change in QOL using EORTC QLQ-BN20 | Baseline to 24 months
  EORTC QLQ-BN 20 consists of 20 items and measures the functioning and symptoms of patients with intracranial malignant disease. Questions can be grouped into 3 multi-item functional scales (visual disorder, motor dysfunction, communication deficit), 7 single items (headaches, seizures, drowsiness, itchy skin, hair loss, weakness of legs and bladder control) and 1 multi-item scale on future uncertainty.
  Scoring is on a scale of 0 to 80, with higher scores indicating worse symptoms. The change score from baseline to 24 months will be calculated by subtracting the 24-month score from the baseline score. Positive values indicate improved symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Minesh Mehta, M.D., Principal Investigator — Miami Cancer Institute at Baptist Health, Inc.; Yazmin Odia, M.D., Principal Investigator — Miami Cancer Institute at Baptist Health, Inc.
Locations (1):
- Miami Cancer Institute at Baptist Health, Inc., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen X, Zhang L, Zhang IY, Liang J, Wang H, Ouyang M, Wu S, da Fonseca ACC, Weng L, Yamamoto Y, Yamamoto H, Natarajan R, Badie B. RAGE expression in tumor-associated macrophages promotes angiogenesis in glioma. Cancer Res. 2014 Dec 15;74(24):7285-7297. doi: 10.1158/0008-5472.CAN-14-1240. Epub 2014 Oct 17. PMID 25326491
- [Background] van Grinsven EE, Nagtegaal SHJ, Verhoeff JJC, van Zandvoort MJE. The Impact of Stereotactic or Whole Brain Radiotherapy on Neurocognitive Functioning in Adult Patients with Brain Metastases: A Systematic Review and Meta-Analysis. Oncol Res Treat. 2021;44(11):622-636. doi: 10.1159/000518848. Epub 2021 Sep 3. PMID 34482312
- [Background] Yang L, Liu Y, Wang Y, Li J, Liu N. Azeliragon ameliorates Alzheimer's disease via the Janus tyrosine kinase and signal transducer and activator of transcription signaling pathway. Clinics (Sao Paulo). 2021 Mar 8;76:e2348. doi: 10.6061/clinics/2021/e2348. eCollection 2021. PMID 33681944
- [Background] Davis HM, Essex AL, Valdez S, Deosthale PJ, Aref MW, Allen MR, Bonetto A, Plotkin LI. Short-term pharmacologic RAGE inhibition differentially affects bone and skeletal muscle in middle-aged mice. Bone. 2019 Jul;124:89-102. doi: 10.1016/j.bone.2019.04.012. Epub 2019 Apr 24. PMID 31028960
- [Background] Riuzzi F, Sorci G, Sagheddu R, Chiappalupi S, Salvadori L, Donato R. RAGE in the pathophysiology of skeletal muscle. J Cachexia Sarcopenia Muscle. 2018 Dec;9(7):1213-1234. doi: 10.1002/jcsm.12350. Epub 2018 Oct 18. PMID 30334619
- [Background] Chiappalupi S, Sorci G, Vukasinovic A, Salvadori L, Sagheddu R, Coletti D, Renga G, Romani L, Donato R, Riuzzi F. Targeting RAGE prevents muscle wasting and prolongs survival in cancer cachexia. J Cachexia Sarcopenia Muscle. 2020 Aug;11(4):929-946. doi: 10.1002/jcsm.12561. Epub 2020 Mar 11. PMID 32159297
- See also: Miami Cancer Institute — http://cancer.baptisthealth.net/